CLINICAL TRIAL: NCT00189358
Title: A Phase II Study of ZD1839 and Tamoxifen in Patients With Epithelial Ovarian Carcinoma, Cancer of the Fallopian Tube or the Peritoneum Refractory to Platinum- and Taxane-based Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AGO Study Group (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGO-OVAR 2.6
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Ovarian Cancer; Cancer of the Fallopian Tube; Peritoneal Cancer
Keywords: cancer; cancer alternative therapies; ovarian cancer; tyrosine kinase inhibitor
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Neoplasms | interventions — Gefitinib; Tamoxifen

INTERVENTIONS:
Drug: ZD1839
Drug: tamoxifen

SUMMARY:
Although initially responsive to cytoreductive surgery and platinum- and/or taxane-based chemotherapy, a majority of patients with epithelial ovarian cancer, cancer of the fallopian tube or the peritoneum will eventually relapse. Recurrence within 6 months after completing platinum-containing chemotherapy indicates a platinum-refractory cancer disease. New therapeutic strategies are required in platinum-refractory disease. Inhibition of growth signals induced by the epidermal growth factor receptor pathway, or by the estrogen receptor pathway provides promising targets in epithelial ovarian cancer, cancer of the fallopian tube or the peritoneum. The trial is to evaluate the safety and tolerability of the combination of the epidermal growth facto tyrosine kinase inhibitor ZD1839 and the clinically established antiestrogen tamoxifen.

ELIGIBILITY:
Inclusion Criteria:

histologically confirmed epithelial ovarian cancer, cancer of the fallopian tube or peritoneum refractory to platinum- and taxane-based chemotherapy measurable or non-measurable disease written informed consent aged 18 years or older Karnofsky performance status > 60%

Exclusion Criteria:

complete bowel obstruction symptomatic brain metastases known hypersensitivity to evaluated drugs inadequate kidney function inadequate hepatic function evidence of clinically active interstitial lung disease history of congestive heart failure > NYHA 2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Safety and tolerability

SECONDARY OUTCOMES:
objective response rate
time to progression
overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Wagner, Prof.Dr., Principal Investigator — AGO Study Group
Locations (1):
- Dept. of Gynecology, Evangelisches Krankenhaus, Düsseldorf, Germany

REFERENCES:
- [Result] Wagner U, du Bois A, Pfisterer J, Huober J, Loibl S, Luck HJ, Sehouli J, Gropp M, Stahle A, Schmalfeldt B, Meier W, Jackisch C; AGO Ovarian Cancer Study Group. Gefitinib in combination with tamoxifen in patients with ovarian cancer refractory or resistant to platinum-taxane based therapy--a phase II trial of the AGO Ovarian Cancer Study Group (AGO-OVAR 2.6). Gynecol Oncol. 2007 Apr;105(1):132-7. doi: 10.1016/j.ygyno.2006.10.053. Epub 2006 Dec 11. PMID 17161453